CLINICAL TRIAL: NCT06285643
Title: A Phase 2, Randomized, Double-blind, Sham Surgery-controlled Study of the Efficacy and Safety of Intraputaminal AAV2-GDNF in the Treatment of Adults With Moderate Stage Parkinson's Disease
Brief Title: A Study of AAV2-GDNF in Adults With Moderate Parkinson's Disease (REGENERATE-PD)
Acronym: REGENERATE-PD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AskBio Inc (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASK-PD5-CS201
Record Dates: First submitted 2024-02-14; First posted 2024-02-29 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Gene therapy
MeSH Terms: conditions — Parkinson Disease | interventions — Biological Products

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AAV2-GDNF (Experimental)
  Interventions: Drug: AAV2-GDNF gene therapy
- Control Surgery (Sham Comparator)
  Interventions: Procedure: control surgery

INTERVENTIONS:
Drug: AAV2-GDNF gene therapy — Bilateral image-guided infusion of AAV2-GDNF into putamen, single dose
  Other Names: Biological
  Arms: AAV2-GDNF
Procedure: control surgery — Bilateral partial burr/twist holes without dural penetration
  Arms: Control Surgery

SUMMARY:
The objective of this randomized, surgically controlled, double-blinded, Phase 2 study is to evaluate the safety and efficacy of AAV2-GDNF delivered to the putamen in subjects with moderate Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

Age

1. Male and female adults 45-75 years of age inclusive, at the time of signing of informed consent Type of Subject and Disease Characteristics
2. Diagnosed with Parkinson's disease in the past 4-10 years (inclusive) as defined by the following:

   1. Presence of bradykinesia PLUS any of the following:

      * Rigidity
      * Rest tremor
      * Postural instability
   2. Presence of motor fluctuations as measured by the PD Motor Diary
   3. Stable anti-parkinsonian medication regimen for >/= 4 weeks prior to screening
   4. Must demonstrate responsiveness to levodopa therapy

Exclusion Criteria:

* Known history or current evidence of medical, genetic, or neurological conditions that may provide an alternative to idiopathic PD diagnosis
* Presence or history of significant vascular and/or cardiovascular disease
* Presence of significant cognitive impairment, poorly controlled depression/anxiety
* Presence or history of psychosis or impulse control disorder
* History of malignancy other than treated cutaneous squamous or basal cell carcinomas
* Presence of clinically relevant conditions that could compromise surgical suitability and/or subject safety
* Contraindication to magnetic resonance imaging and/or use gadolinium-based contrast agents
* Prior history of brain surgery including, but no limited: DBS, pallidotomy focused ultrasound thalamotomy, or other experimental neurosurgical procedure
* Chronic immunosuppressive therapy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Month 18 on PD Motor Diary | 18 months
  Normalized Good ON time per Hauser Diary

CONTACTS AND LOCATIONS:
Locations (39):
- United States (27):
  - UCI Alpha Clinic (Neurology), Irvine, California
  - Loma Linda University (Neurology), Loma Linda, California
  - Loma Linda University (Surgical), Loma Linda, California
  - University of California San Francisco (Neurology), San Francisco, California
  - University of San Francisco (Surgical), San Francisco, California
  - CenExel Rocky Mountain Clinical Research (Neurology), Englewood, Colorado
  - Georgetown University (Neurology), Washington D.C., District of Columbia
  - Parkinson's Disease and Movement Disorders Center of Boca Raton (Neurology), Boca Raton, Florida
  - Parkinson's Disease Treatment Center of Southwest Florida (Neurology), Port Charlotte, Florida
  - Emory University (Surgical), Atlanta, Georgia
  - Rush University Medical Center (Neurology), Chicago, Illinois
  - University of Kansas Medical Center (Neurology), Kansas City, Kansas
  - Massachusetts General Hospital (Neurology), Boston, Massachusetts
  - Massachusetts General Hospital (Surgical), Boston, Massachusetts
  - Michigan State University (Neurology), East Lansing, Michigan
  - Quest Research Institute (Neurology), Farmington Hills, Michigan
  - Cleveland Clinic Lou Ruvo (Neurology), Las Vegas, Nevada
  - University of North Carolina (Neurology), Chapel Hill, North Carolina
  - Duke Neurosurgery (Surgical), Durham, North Carolina
  - Duke University (Neurology), Durham, North Carolina
  - Ohio State University (Surgical), Columbus, Ohio
  - University of Pennsylvania (Neurology), Philadelphia, Pennsylvania
  - Vanderbilt University (Neurology), Nashville, Tennessee
  - Houston Methodist (Neurology), Houston, Texas
  - Houston Methodist (Surgical), Houston, Texas
  - EvergreenHealth Research Department (Neurology), Kirkland, Washington
  - University of Wisconsin (Neurology), Madison, Wisconsin
- Germany (5):
  - Charité - Universitätsmedizin Berlin (Surgical), Berlin
  - Philipps-Universität Marburg (Neurology), Marburg
  - Universitätsklinikum Tübingen (Neurology), Tübingen
  - Universitätsklinikum Tübingen (Surgical), Tübingen
  - Universitätsklinikum Würzburg (Neurology), Würzburg
- Poland (5):
  - Copernicus Podmiot Leczniczy, Szpital św. Wojciecha (Neurology), Gdansk
  - Specjalistyczna Praktyka Lekarska Prof. Grzegorz Opala (Neurology), Katowice
  - Mazowiecki Szpital Bródnowski (Neurology), Warsaw
  - Mazowiecki Szpital Bródnowski (Surgical), Warsaw
  - Samodzielny Publiczny Szpital Kliniczny im. Prof. W. Orłowskiego CMKP (Neurology), Warsaw
- United Kingdom (2):
  - North Bristol NHS Trust - Southmead Hospital (Neurology), Bristol
  - University Hospital of Wales (Surgical), Cardiff

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Nurse Navigator Service for Potential Participants — https://mytomorrows.com/ask-bio/regenerate-pd/en-us/